CLINICAL TRIAL: NCT01072890
Title: Phase I Study of the Combination of Temsirolimus (CCI-779) and Pazopanib (GW786034) in Patients With Advanced Solid Tumors
Brief Title: Temsirolimus and Pazopanib in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: GlaxoSmithKline (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200917514; UCDCC#222 (Other: University of California Davis)
Record Dates: First submitted 2010-02-16; First posted 2010-02-22 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Solid Tumors
Keywords: Temsirolimus, Pazopanib
MeSH Terms: interventions — temsirolimus; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus and Pazopanib (Experimental)
  Interventions: Drug: Temsirolimus, Pazopanib

INTERVENTIONS:
Drug: Temsirolimus, Pazopanib — Patients will be treated on an outpatient basis with both temsirolimus and pazopanib. All patients will receive temsirolimus intravenously (IV) weekly days 1, 8, 15, and 22. Patients will receive oral pazopanib on a daily basis starting day 1. Treatment will be administered on 28 day cycles. Patients will be in this study for a minimum of 8 weeks or 2 cycles.
  Other Names: Torisel; Votrient

SUMMARY:
The purpose of this study is to test the safety of temsirolimus and pazopanib at different doses. Patients who have an advanced cancer that is not felt to benefit from standard treatment or are no longer responding to other treatment will be asked to take part in this study. The study hypothesis is that temsirolimus and pazopanib can be administered safely in combination and that combined targeting of the mammalian target of rapamycin (mTOR) and vascular endothelial growth factor receptor (VEGFR) signaling pathways will be effective in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
Despite encouraging clinical activity reported with single-agent VEGF inhibitors, mTOR inhibitors, and other novel agents, patients rarely achieve complete disease response and ultimately undergo disease progression. The limited efficacy of single-target inhibition may be due to numerous, overlapping signaling pathways involved in Renal Cell Carcinoma proliferation and growth. A strategy of multi-target "vertical inhibition" of the overlapping aberrant VEGF and mTOR pathways by combination therapy may translate to enhanced efficacy over each single agent alone. We hypothesize that temsirolimus and pazopanib can be administered safely in combination and that combined targeting of the mTOR and VEGFR signaling pathways will be effective in treating patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective.
* Age ≥ 18 years old
* Zubrod (ECOG) Performance Status 0 - 2
* May have measurable or non-measurable disease.
* Adequate bone marrow and organ function as assessed by the following within 14 days prior to registration.
* Any number of prior chemotherapy regimens is allowed.
* Any prior chemotherapy, immunotherapy or targeted therapy must have been completed at least 2 weeks prior to start of this protocol and all side effects (except alopecia, lymphopenia and hyperglycemia) resolved to grade 1 or less. Any prior radiation must have been completed at least 2 weeks prior to start of therapy.
* Pregnant or nursing women are ineligible because of the risk to the fetus. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.
* Ability to swallow and retain oral medications.

Exclusion Criteria:

* Prior treatment with an mTOR inhibitor or pazopanib.
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Symptomatic or uncontrolled brain metastasis.
* Must have a EKG within 14 days of registration and a QTc of < 480 msec. If the initial QTc is > 480 msec, two subsequent EKGs should be obtained within 5 minutes.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C due to the immunosuppressive effects of temsirolimus.
* Active clinically serious infection > CTCAE Grade 2.
* Fasting cholesterol > 350mg/dL and fasting triglycerides > 400mg/dL
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy. Therapeutic anticoagulation with warfarin, heparin or low molecular weight heparin is not allowed. Patients may not have had an arterial thrombotic event within the past 6 months.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug.
* May not take known strong CYP3A4 inducers such as rifampin or St. John's wort or strong CYP3A4 inhibitors such as ketoconazole, diltiazem, or verapamil.
* Known or suspected allergy to temsirolimus or pazopanib, any similar agents such as the rapamycin analog sirolimus, or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of temsirolimus and pazopanib when given in combination to patients with advanced solid tumors. | Every 4 weeks (Cycle)

SECONDARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of temsirolimus and pazopanib when given in combination to patients with advanced solid tumors and to recommend a phase II dose for the combination. | Every 4 weeks (Cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N Lara, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Derived] Semrad TJ, Eddings C, Dutia MP, Christensen S, Lara PN Jr. Phase I study of the combination of temsirolimus and pazopanib in advanced solid tumors. Anticancer Drugs. 2013 Jul;24(6):636-40. doi: 10.1097/CAD.0b013e3283618b7b. PMID 23698253
- See also: University of California Davis Cancer Center — http://www.ucdmc.ucdavis.edu/CANCER/